CLINICAL TRIAL: NCT00690963
Title: A Phase I/II Dose Escalation Trial Using Hypofractionation With Individualized Differential Boosting With Respiratory Gated Intensity-modulated Radiation Therapy (IMRT) in the Treatment of Non-small Cell Lung Cancer.
Brief Title: Individual Boosting in Non-Small Cell Lung Cancer Using Hypofractionation, Intensity-modulated Radiation Therapy and Respiratory Gating
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: AHS Cancer Control Alberta (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LU-24123
Record Dates: First submitted 2008-06-03; First posted 2008-06-05 (Estimated); Last update posted 2016-04-06 (Estimated); Status verified 2016-04

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: Radiotherapy; Intensity-Modulated; Dose Fractionation
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Radiotherapy — Dose excalation based on normal tissue toxicity using 5 dose bins ranging from 56.8 Gy/ 27 fractions to 67.3 Gy in 27 fractions.

SUMMARY:
Patients who have inoperable non-small cell lung cancer are presently treated with chemotherapy and radiation therapy. Despite this combined approach, the vast majority of patients will have their cancer recur after treatment. A recurrence is not curable at this time. Because of the sensitivity of surrounding structures to chest irradiation, it has not been possible to give radiation doses that can cure many of these tumors. Intensity-modulated radiation therapy is a special form of radiotherapy delivery that allows doctors to reduce the amount of radiation dose to normal tissues and therefore reduce side effects. The reduction of radiation side effects may allow more radiation to be delivered to tumors, therefore improving tumor control and possibly longevity of patients. The purpose of this study is to determine whether the combination of custom designed intensity-modulated radiotherapy (based on individual tumor anatomy) with regular chemotherapy, will be safe enough to allow further intensification of radiation treatment.

DETAILED DESCRIPTION:
All patients must have a satisfactory IMRT plan prior to starting radiation therapy, which will commence concurrently with chemotherapy. All patients will be treated to a minimum of 48 Gy in 20 daily fractions over 4 weeks [2.4 Gy per fraction (fx)], to the planning target volume (PTV) defined by pre chemotherapy CT with PET imaging. This is approximately biologically equivalent to a dose of 54 Gy in 27# (5 fractions/week). A differential boosting will then be selected from one of 5 dose escalation schemes. The total individual radiotherapy dose will be prescribed according to the highest dose level that can satisfy all of the set radiotherapy planning constraints for the individual's anatomy. The trial will proceed in 2 phases. In the first phase only the first 3 dose escalation schedules will be used. Once all of these 3 schedules have been deemed safe then dose levels 4 and 5 will be opened up to participation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically-proven, by biopsy or cytology, unresected lung cancer of the following histologic types: Squamous cell carcinoma, Adenocarcinoma, Undifferentiated large cell carcinoma, Non-Small cee; not otherwise specified (NOS, diagnosis on cytology alone)
* Patients with AJCC Stage II, IIIA or IIIB if all detectable tumour can be encompassed by radiation therapy fields, including both the primary tumor and the involved regional lymph nodes
* Patient must be deemed to be suitable to undergo definitive chemo-radiotherapy by the treating Physician.
* Age > = 18
* ECOG/Zubrod status 0-1
* Patients must have measurable disease on CT imaging
* Satisfactory granulocytes, platelets, bilirubin, AST and calculated creatinine clearance
* Dose volume constraints must be met
* Patient must be able to use the breath-held technique

Exclusion Criteria:

* Patients who have undergone complete or subtotal tumour resection
* Patients with post-resection intrathoracic tumour recurrence
* Patients eligible for definitive surgery
* Evidence of any small cell histology
* Prior or concurrent malignancy except non-melanomatous skin cancer unless disease-free for at least 5 years
* Exudative pleural effusion, or pleural effusions with positive cytology. Minimal pleural effusions which are too small to safely tap (i.e. not visible on chest x-ray) are eligible.
* Patients with myocardial infarction within the preceding 6 months or symptomatic heart disease, including angina, congestive heart failure and uncontrolled arrhythmias
* Pregnant women are ineligible. Patients with childbearing potential must practice appropriate contraception
* Patients with FEV1 <= 0.8. Patients with FEV1 >0.8 and <1.0 to be discussed with a Respiratory Physician

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2008-09; Primary Completion 2016-09 (Estimated); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
Toxicity of treatment | 90 days (Acute), 5 years (Late)

SECONDARY OUTCOMES:
Local control | 5 years
overall survival | 5 years
Disease Free Survival | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Wilson Roa, MSc, MD, FRCPC, Study Chair — Cross Cancer Institute, Alberta Health Services
Locations (1):
- Cross Cancer Institute, Edmonton, Alberta, Canada